CLINICAL TRIAL: NCT00232544
Title: RCT of a Telecommunications System in Sleep Apnea
Brief Title: Telecommunications System in Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IIR 02-230
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Results first posted 2014-02-17 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-09

CONDITIONS: Sleep Apnea, Obstructive
Keywords: sleep apnea, obstructive; Quality of Life; Depression; Patient Compliance
MeSH Terms: conditions — Sleep Apnea, Obstructive; Depression; Patient Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TLC-CPAP (Experimental): A telephone-linked communication (TLC) system for promoting adherence to continuous positive airway pressure (CPAP)
  Interventions: Device: Telecommunications system
- TLC-Control (Placebo Comparator): A TLC system for providing general health education
  Interventions: Other: TLC-Control

INTERVENTIONS:
Device: Telecommunications system — The telecommunications system is designed to improve patient adherence with prescribed positive airway pressure.
  Arms: TLC-CPAP
Other: TLC-Control — A TLC system for providing general health education
  Arms: TLC-Control

SUMMARY:
This study is investigating the effects of a telecommunications system designed to improve patient adherence with prescribed positive airway pressure (CPAP).

DETAILED DESCRIPTION:
Background/Rationale:

Obstructive sleep apnea syndrome (OSAS) is an important chronic disease of adults, affecting an estimated 4% of men and 2% of women in the United States. Nasal continuous positive airway pressure (CPAP) has been demonstrated to ameliorate the symptoms and neurobehavioral consequences of OSAS. Unfortunately, patient adherence with prescribed CPAP is low, diminishing the benefits obtained from this expensive therapy. Nurse-administered patient education and monitoring of CPAP use through home visits has been shown to be effective in significantly improving CPAP adherence. Given the logistic complexity of delivering this service and its costs, it is unlikely to be disseminated widely into clinical practice. An alternative, using advanced telecommunications technology to deliver similar adherence improvement services, is proposed for study.

Objective(s):

Use of telecommunications systems with other important health-related behaviors such as medication-taking, diet, and exercise have demonstrated significant improvements in therapy adherence.

Methods:

This research project represents a randomized controlled trial of a Telephone-Linked Communications (TLC) system designed to improve CPAP adherence (TLC-CPAP). The study will enroll adults with OSAS who are being started on nasal CPAP therapy. Subjects will be randomized to TLC-CPAP or an attention placebo control group. The effect of TLC on CPAP use and on disease-specific quality of life (QOL), OSAS-related symptoms, depression, and vigilance over a 12-month interval will be assessed.

The intervention and control groups will be compared to assess differences in potential confounders including age, sex, OSAS severity, CPAP pressure level, comorbid illness, physician specialty status, BMI, socioeconomic status, and marital status. Each of the outcome variables (all of which are continuous variables) will be compared between intervention and control groups using multivariate analyses to adjust for any potential confounders that differ between groups. Multivariate models will include appropriate tests of interactions. All analyses will be performed using an intent-to-treat approach.

Status:

Completed

Impact:

This Telephone-Linked Communications (TLC) technology offers an effective, low-cost, and easy-to-use means of providing disease-specific education, monitoring, and counseling to improve adherence with therapy.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of obstructive sleep apnea syndrome plus polysomnography demonstrating greater than 10 apneas plus hypopneas per hour of sleep
* Age 18-80 years
* Ability to use a telephone without assistance

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2004-10; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David William Sparrow, DSc, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Sparrow D, Aloia M, Demolles DA, Gottlieb DJ. A telemedicine intervention to improve adherence to continuous positive airway pressure: a randomised controlled trial. Thorax. 2010 Dec;65(12):1061-6. doi: 10.1136/thx.2009.133215. Epub 2010 Sep 29. PMID 20880872

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TLC-CPAP | TLC-Control
Started | 124 | 126
Completed | 104 | 111
Not Completed | 20 | 15
Not completed — Lost to Follow-up | 20 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TLC-CPAP | TLC-Control | Total
Number analyzed (Participants) | 124 | 126 | 250
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 56 [48 to 63] | 54 [45 to 62] | 55 [46 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 21 | 45
  Male | 100 | 105 | 205
Region of Enrollment [Number; unit: participants]
  United States | 124 | 126 | 250

OUTCOME MEASURES:

1. Primary Outcome: Objective CPAP Use
Description: Mean nightly hours of CPAP use over 12 months
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: log(hours/night)
Arm/Group | TLC-CPAP | TLC-Control
Number analyzed (Participants) | 104 | 111
log(hours/night) | 0.437 [0.165 to 0.708] | -0.066 [-0.376 to 0.243]

2. Secondary Outcome: Daytime Vigilance
Description: A measure of behavioral alertness. Specifically the metric we used was the mean reaction time, the time it took for a subject to respond to a visual stimulus (light displayed on a screen at random intervals) by hitting a button.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: ms
Arm/Group | TLC-CPAP | TLC-Control
Number analyzed (Participants) | 104 | 111
ms | 293.7 [279.9 to 307.6] | 324.0 [302.2 to 345.8]

ADVERSE EVENTS:
Arm/Group | TLC-CPAP | TLC-Control
Serious Adverse Events (participants affected / at risk) | 1/124 | 0/126
Other Adverse Events (participants affected / at risk) | 0/124 | 0/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TLC-CPAP (N=124) | TLC-Control (N=126)
Death (Gastrointestinal disorders) | 1 (1) | 0 (0) — Patient died in hospital while being treated for bowel obstruction. PI and IRB concluded death not study related.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes